CLINICAL TRIAL: NCT01070745
Title: Ibuprofen vs. Indomethacin as Second Course of Therapy for Resistant PDA in Low Birth Weight Neonates
Brief Title: Second Course of Therapy for Resistant Patent Ductus Arteriosus (PDA)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes in approach to PDA therapy
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Cathy Hammerman, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chammerman3
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2010-02

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Indomethacin; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin; Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin for resistant PDA (Experimental): Treatment with second course of indomethacin
  Interventions: Drug: Indomethacin
- Ibuprofen for resistant PDA (Experimental): Ibuprofen as second course of therapy
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Indomethacin — Three doses of intravenous (IV) indomethacin at 0.2 mg/kg/dose given over 30 minutes, at intervals of 12 hours
  Other Names: Indomed
  Arms: Indomethacin for resistant PDA
Drug: Ibuprofen — 10 mg/kg infused over 30 minutes, followed by two doses of 5mg/kg each at 24 hour intervals
  Other Names: Arfen
  Arms: Ibuprofen for resistant PDA

SUMMARY:
Patency of the ductus arteriosus (PDA) is functionally essential for fetal circulation, however persistence of ductal patency postnatally may have significant adverse hemodynamic effects in the neonate. Medical therapy for PDA predominantly involves the administration of one of two non-steroidal anti-inflammatory drugs: indomethacin or ibuprofen. Both of these therapies have been shown to be successful in mediating ductal closure in approximately 70% of treated infants.

However, the need for a second course of treatment for PDA closure remains quite common. The investigators hypothesize that, because of small differences between the two drugs, a greater percentage of infants who did not respond to a first course of therapy with indomethacin will respond to a second course with ibuprofen than to a repeat course of indomethacin.

As such, the investigators aim to compare secondary therapy with a repeat course of indomethacin to secondary therapy with ibuprofen in infants whose ductus remained patent after a first course of therapy with indomethacin.

ELIGIBILITY:
Inclusion Criteria:

* Inborn premature neonates (birth weight [BW] <1500 grams) being treated in the neonatal intensive care unit of the Shaare Zedek Medical Center and diagnosed as still having a hemodynamically significant patent ductus arteriosus (hsPDA) after a first course of therapy with indomethacin, will be considered as potential candidates for study pending response to initial therapy and pending parental consent.

Exclusion Criteria:

* Any baby not considered viable
* Any baby with intraventricular hemorrhage (IVH) grade 3-4 of recent onset (within 3 days). [If no head ultrasound has been performed within the last 3-4 days, one should be performed prior to onset of study.]
* Any baby with dysmorphic features or congenital abnormalities
* Any baby with structural heart disease other than PDA
* Any baby with documented infection,
* Any baby with thrombocytopenia (<50,000).

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in ductal closure rates in those infants who do not respond to a first course of therapy | 2.5 years

SECONDARY OUTCOMES:
More infants who did not respond to a first course of therapy with indomethacin who respond to a second course with ibuprofen than to a repeat course of indomethacin | 2.5 years
Secondary treatment with ibuprofen, as opposed to indomethacin, will not be associated with increased side effects | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Investigator
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel